CLINICAL TRIAL: NCT01606709
Title: A Prospective Comparison of Transcriptional Profiling of Luteal Phase Endometrial Biopsies After Induction of Oocyte Maturation With a Gonadotropin Releasing Hormone (GnRH) Agonist or Human Chorionic Gonadotropins (hCG)
Brief Title: Gene Expression Profile After Gonadotropin Releasing Hormone (GnRH) Agonist Trigger of Oocyte Maturation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult to recruit patients
Sponsor: UConn Health (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Lawrence Engmann, MD, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11-168-1
Record Dates: First submitted 2012-05-19; First posted 2012-05-28 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Endometrial Receptivity; Ovarian Hyperstimulation Syndrome
Keywords: GnRHa trigger; endometrial gene profile; quality of life
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Gonadotropin-Releasing Hormone; Leuprolide; Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GnRH agonist trigger (Experimental): Induction of oocyte maturation with GnRH agonist
  Interventions: Drug: GnRH agonist
- hCG trigger (Active Comparator): Induction of oocyte maturation with hCG
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: GnRH agonist — GnRH agonist 1mg one dose
  Other Names: leuprolide acetate,; lupron
  Arms: GnRH agonist trigger
Drug: hCG — 5,000 IU one dose
  Other Names: Pregnyl
  Arms: hCG trigger

SUMMARY:
The purpose of this study is to compare gene expression profiles in endometrial biopsies during the window of implantation after triggers of oocyte maturation using GnRH agonist or hCG and compared with their natural cycles in order to identify genes that may be dysregulated in GnRH agonist-triggered cycles.

The investigators also intend to evaluate patients feeling of well being and physical quality of life after GnRH agonist trigger compared with hCG trigger.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome (OHSS) is an iatrogenic complication of controlled ovarian hyperstimulation (COH) which may result in significant morbidity and rarely mortality as well as significant financial and psychological distress. The use of a GnRH agonist for induction of final oocyte maturation in ovarian stimulation cycles utilizing GnRH antagonist for pituitary suppression has proven to be an effective method of preventing the risk of OHSS development.

Unfortunately, some studies, but not all, have also reported lower pregnancy rates in these cycles as compared to cycles using hCG trigger and this has been attributed to possible impaired endometrial receptivity.

The investigators intend to obtain endometrial biopsies collected from the same subject in a natural cycle and then a biopsy during either a GnRH agonist or hCG triggered stimulation. Expression profiles of mRNAs will first be screened using microarray technology. Relative levels of specific mRNAs that display altered expression in the GnRH-triggered samples, as assayed by microarray, will then be confirmed by real-time, quantitative reverse transcription/polymerase chain reaction (Q-PCR). The investigators shall also evaluate patients feeling of well being and physical quality of life after GnRH agonist trigger compared with hCG trigger.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donors
* Ages between 21 and 33
* Normal baseline serum FSH < 10mIU/mL

Exclusion Criteria:

* Hypothalamic dysfunction
* Smokers
* Baseline serum FSH ≥ 10mIU/mL

Ages: 21 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Engmann, MD, MRCOG, Principal Investigator — UConn Health
Locations (1):
- UCHC Division of Reproductive Endocrinology, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GnRH Agonist Trigger | hCG Trigger
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GnRH Agonist Trigger | hCG Trigger | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Endometrial Gene Expression Profile
Description: Microarray of gene expression in the midluteal phase
Time Frame: 7 days after trigger of oocyte maturation
Population: Inadequate RNA quality to completely analyze gene expression
Arm/Group | GnRH Agonist Trigger | hCG Trigger
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Life Survey After Ovarian Stimulation and GnRHa or hCG Trigger
Time Frame: At baseline and up to 7 days after trigger of oocyte maturation
Population: Too few patients completed survey to meaningfully analyze data
Arm/Group | GnRH Agonist Trigger | hCG Trigger
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 weeks for each patient
Arm/Group | GnRH Agonist Trigger | hCG Trigger
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No